CLINICAL TRIAL: NCT03863834
Title: Clinical Evaluation of Safety and Efficacy of Radio-Frequency Assisted Lipolysis (RFAL) of Breast Envelope and Nipple-Areolar Complex (NAC) Position
Brief Title: Clinical Evaluation of RFAL of Breast Envelope and NAC Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0607738
Record Dates: First submitted 2019-02-27; First posted 2019-03-05 (Actual); Results first posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2021-02

CONDITIONS: Breast Lift

STUDY DESIGN:
Intervention Model Description: Subjects will receive the treatment and outcome will be followed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment arm (Experimental): Subjects receive the RFAL treatment
  Interventions: Device: InModeRF

INTERVENTIONS:
Device: InModeRF — InModeRF minimally invasive treatment based on Radiofrequency-assisted lipolysis (RFAL) technology

SUMMARY:
This single center clinical study is intended to determine the safety and efficacy of using Radiofrequency (RF) energy for minimally invasive breast lift procedure.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of RFAL for the Breast Envelope and Nipple-Areolar Complex (NAC) Position as measured by Vectra 3D circumferential imaging system (Canfield, NJ)

ELIGIBILITY:
Inclusion Criteria:

* Informed consent agreement signed by the subject.
* Healthy females 21 to 60 years of age.
* Presence of grade I-III Breast Ptosis, mastopexy with history of breast augmentation, correction of asymmetry, mastopexy alone, mastopexy following implant removal and modest breast reduction in combination with or without lipoaspiration.
* Post-menopausal or surgically sterilized or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study (i.e., oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide, or abstinence).
* Willingness to follow the treatment and follow-up schedule and the post-treatment care.
* All participants must have a recorded mammogram before the beginning of the study.

Exclusion Criteria:

* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body.
* Permanent implant in the treated area such as metal plates and screws, silicone implants or an injected chemical substance.
* Current or history of skin cancer (remission of 5 years), or current condition of any other type of cancer, or pre-malignant moles.
* Severe concurrent conditions, such as cardiac disorders, epilepsy, uncontrolled hypertension, and liver or kidney diseases.
* History of bleeding coagulopathies or use of anticoagulants in the last 2 weeks.
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV or use of immunosuppressive medications.
* Poorly controlled endocrine disorders, such as diabetes or thyroid dysfunction.
* Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
* Significant systemic illness or occult systemic illness.
* Illness, infection or skin diseases localized in area of treatment.
* Other therapies or medication which may interfere with treatment.
* Breastfeeding, pregnant, or planning to become pregnant during the study.
* Allergy to lidocaine or other anaesthesia.
* Recent surgery in treatment area within the past 6 months.
* Participation in a study of another device or drug within 3 months prior to enrolment or during this study.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the patient to participate in this study.
* As per the practitioner's discretion, refrain from treating any condition that might make it unsafe for the patient.

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-13 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Unger, MD, Principal Investigator — Maxwell Aesthetics 2020 21st Ave, South, Nashville, TN, 37212, USA
Locations (1):
- Jacob G Unger MD, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm
Started | 12
Completed | 9
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Only subjects that finished 12 month follow up were analyzed
Arm/Group | Treatment Arm
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Sternal Notch to Left Nipple Distance in centimeters [Mean (Standard Deviation); unit: centimeters] — static measurements in cm of distance from sternal notch to nipple
  centimeters | 24.56 (1.88)
sternal notch to right nipple distance in cm [Mean (Standard Deviation); unit: centimeters] | 25.25 (2.20)
right nipple to im crease [Mean (Standard Deviation); unit: centimeters] | 11.44 (3.18)
left nipple to crease [Mean (Standard Deviation); unit: centimeters] | 12.44 (3)
right base width [Mean (Standard Deviation); unit: centimeters] | 12.93 (1.76)
left base width [Mean (Standard Deviation); unit: centimeters] | 13.29 (2.14)
nipple to nipple [Mean (Standard Deviation); unit: centimeters] | 21.63 (1.71)

OUTCOME MEASURES:

1. Primary Outcome: Measurements of Distance (cm) Between Breast Area Reference Points (Nipple to Nipple)
Description: Regular and 3D Vectra photos will be taken at all time points.
  Additional evaluation of changes in breast shape, including upper pole fullness, breast projection, and bottoming out will be assessed by static measurements (cm) of:
  * Sternal Notch to Nipple
  * Nipple to Inframammary Fold (IMF)
  * Base Width (at point of breast take off from chest wall)
  * Nipple to nipple
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Treatment Arm
Number analyzed (Participants) | 9
centimeters | 20.6 (1.35)

2. Primary Outcome: Number of Adverse Events Will be Assessed Based on Frequency, Severity and Causality Data.
Description: Safety will be evaluated by observation, assessment and recording of adverse events, if occur. Evaluations will be done immediately after treatment and at all follow-up visits. Each occurrence will be described in a table presenting data including severity (mild, moderate or severe), causality (relationship to the device or the treatment), treatment and resolution. Data will be summarized and adverse event significance will be considered based on combination of the above listed items.
Time Frame: 12 months
Measure: Number; unit: number of events
Arm/Group | Treatment Arm
Number analyzed (Participants) | 9
number of events | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT03863834/Prot_SAP_000.pdf